CLINICAL TRIAL: NCT04537494
Title: PREVENT: PRobiotics for EVEry Newborn vs Treatment-as-Needed Comparative Effectiveness Trial
Brief Title: PRobiotics for EVEry Newborn Trial
Acronym: PREVENT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The Hospital for Sick Children (Other)
Responsible Party: Principal Investigator, Patricia Parkin, Professor, Senior Associate Scientist, Staff Pediatrician, The Hospital for Sick Children
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 1000064700
Record Dates: First submitted 2020-01-27; First posted 2020-09-03 (Actual); Last update posted 2025-05-18 (Actual); Status verified 2025-05

CONDITIONS: Colic; Infantile
Keywords: Colic; Probiotic; Infant
MeSH Terms: conditions — Colic

STUDY DESIGN:
Masking Description: For the 2 Randomized arms, all parties were masked. For the 2 Parent Preference arms, all parties were unmasked (open label)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- Prevention (Randomized) (Active Comparator): Oral supplementation with the probiotic L. reuteri administered to every newborn within the first week of life for 12 weeks
  Interventions: Dietary Supplement: L. reuteri
- Treatment-as-needed (Randomized) (Other): Supplementation with the probiotic L. reuteri after randomization, to infants who develop excessive cry/fuss up to 12 weeks of age
  Interventions: Dietary Supplement: L. reuteri
- Prevention (Parent Preference) (Active Comparator): Oral supplementation with the probiotic L. reuteri administered to every newborn within the first week of life for 12 weeks
  Interventions: Dietary Supplement: L. reuteri
- Treatment-as-needed (Parent Preference) (Other): Supplementation with the probiotic L. reuteri after randomization, to infants who develop excessive cry/fuss up to 12 weeks of age
  Interventions: Dietary Supplement: L. reuteri

INTERVENTIONS:
Dietary Supplement: L. reuteri — Probiotic
  Other Names: BioGaia

SUMMARY:
The aim of the study is to compare prevention (oral supplementation with the probiotic L. reuteri administered to every newborn within the first week of life for 12 weeks) with treatment-as-needed (supplementation with the probiotic L. reuteri after randomization, to infants who develop excessive cry/fuss up to 12 weeks of age). This is a single site pilot study to assess feasibility for a full trial.

DETAILED DESCRIPTION:
One in five infants experience colic, defined as recurrent and prolonged episodes of crying and fussing with no obvious cause in healthy infants less than 5 months of age. There is evidence to support the role of the probiotic L. reuteri for treatment of colic in breastfed babies and for prevention of colic. However, these two options (prevention vs treatment-as-needed) have not been previously compared head-to-head. The study aims determine if oral supplementation with the probiotic L. reuteri administered to every newborn within the first week of life for 12 weeks (prevention) is superior to treatment-as-needed, as measured by daily cry/fuss duration at 6 and 12 weeks of age.

ELIGIBILITY:
Inclusion Criteria:

1. 1 to 7 days of age
2. term (37 to 41 weeks)
3. breast or formula fed
4. birth weight > 2500 grams
5. parental consent

Exclusion Criteria:

1. congenital or other medical disorders
2. parents unable to communicate in English or French

Ages: 1 Day to 7 Days | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 32 (Actual)
Dates: Start 2021-12-01 (Actual); Primary Completion 2023-09-08 (Actual); Study Completion 2023-09-08 (Actual)

PRIMARY OUTCOMES:
Combined infant daily cry/fuss duration | Baseline
  The primary outcome will be infant daily cry/fuss duration (combined cry and fuss in minutes) measured using the modified Baby's Day Diary over a 48 hour period.
Combined infant daily cry/fuss duration | 6 weeks
  The primary outcome will be infant daily cry/fuss duration (combined cry and fuss in minutes) measured using the modified Baby's Day Diary over a 48 hour period.
Combined infant daily cry/fuss duration | 12 weeks
  The primary outcome will be infant daily cry/fuss duration (combined cry and fuss in minutes) measured using the modified Baby's Day Diary over a 48 hour period.

SECONDARY OUTCOMES:
Infant daily cry duration | Baseline
  Daily cry duration will be examined separately
Infant daily cry duration | 6 weeks
  Daily cry duration will be examined separately
Infant daily cry duration | 12 weeks
  Daily cry duration will be examined separately
Infant daily fuss duration | Baseline, 6 and 12 weeks of age
  Daily fuss duration will be examined separately
Infant daily fuss duration | Baseline
  Daily fuss duration will be examined separately
Infant daily fuss duration | 6 weeks
  Daily fuss duration will be examined separately
Infant colic | 12 weeks
  Daily cry/fuss of at least 180 minutes
Infant daily sleep duration | Baseline
  Sleep duration will be measured objectively using actigraphy worn around the infant's ankle over a sock.
Infant daily sleep duration | 6 weeks
  Sleep duration will be measured objectively using actigraphy worn around the infant's ankle over a sock.
Infant daily sleep duration | 12 weeks
  Sleep duration will be measured objectively using actigraphy worn around the infant's ankle over a sock.
Parent (female and male) mental health | Baseline
  Mental health will be measured using the Edinburgh Postnatal Depression Scale, a validated 10-item screening questionnaire. Scores range between 0 and 30 and higher scores mean worse outcome.
Parent (female and male) mental health | 6 weeks
  Mental health will be measured using the Edinburgh Postnatal Depression Scale, a validated 10-item screening questionnaire. Scores range between 0 and 30 and higher score means worse outcome.
Parent (female and male) mental health | 12 weeks
  Mental health will be measured using the Edinburgh Postnatal Depression Scale, a validated 10-item screening questionnaire. Scoring is between o and 30 and higher score means worse outcome.
Parent (female and male) fatigue | Baseline
  Fatigue will be measured using a validated Fatigue Visual Analogue Scale. Scores will range between 0 and 180, higher score means worse outcome
Parent (female and male) fatigue | 6 weeks
  Fatigue will be measured using a validated Fatigue Visual Analogue Scale. Scores will range between 0 and 180, higher score means worse outcome.
Parent (female and male) fatigue | 12 weeks
  Fatigue will be measured using a validated Fatigue Visual Analogue Scale. Scores will range between 0 and 180, higher score means worse outcome
Gut microbial composition, diversity and function | Baseline
  Microbial composition, diversity and function will be measured in infant fecal samples.
Gut microbial composition, diversity and function | 6 weeks
  Microbial composition, diversity and function will be measured in infant fecal samples.
Gut microbial composition, diversity and function | 12 weeks
  Microbial composition, diversity and function will be measured in infant fecal samples.
Adverse effects - digestive upset | 8 weeks
  Number of participants with occurrences of digestive upset (e.g., diarrhea), in the Baby's Day Diary
Adverse effects - digestive upset | 16 weeks
  Number of participants with occurrences of digestive upset (e.g., diarrhea), in the Baby's Day Diary
Adverse effects - growth/length | 8 weeks
  Infant growth (length) will be measured at scheduled health supervision visits
Adverse effects - growth/weight | 8 weeks
  Infant growth (weight) will be measured at scheduled health supervision visits
Adverse effects - growth/head circumference | 8 weeks
  Infant growth (head circumference) will be measured at scheduled health supervision visits
Adverse effects - growth/length | 16 weeks
  Infant growth (length) will be measured at scheduled health supervision visits
Adverse effects - growth/weight | 16 weeks
  Infant growth (weight) will be measured at scheduled health supervision visits
Adverse effects - growth/head circumference | 16 weeks
  Infant growth (head circumference) will be measured at scheduled health supervision visits
Health services utilization | Baseline
  Frequency of assessments
Health services utilization | 6 weeks
  Frequency of assessments
Health services utilization | 12 weeks
  Frequency of assessments

CONTACTS AND LOCATIONS:
Overall Officials: Patricia Parkin, MD, Principal Investigator — The Hospital for Sick Children; Patricia Li, MD, Principal Investigator — The Research Institute of the McGill University Health Centre
Locations (1):
- The Hospital for Sick Children, Toronto, Ontario, Canada